CLINICAL TRIAL: NCT04262700
Title: Customer Outcomes & Value Experiencing A New Monitoring Technology
Acronym: CONVERT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LifeScan Scotland Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FILE-PROT-005120
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention 01 (Experimental): Subjects use new LifeScan provided BGMS for 12 weeks.
  Interventions: Device: LifeScan's new BGMS

INTERVENTIONS:
Device: LifeScan's new BGMS — LifeScan new Blood Glucose Monitoring System (BGMS)

SUMMARY:
To investigate whether novel insight features in new Blood Glucose Monitoring System (BGMs) can improve glycemic control.

ELIGIBILITY:
Inclusion Criteria Summary:

* Diagnosed with Type 1 diabetes mellitus or Type 2 diabetes mellitus for ≥ 3 month prior to screening
* Currently performing self-monitoring of blood glucose (SMBG) at home for diabetes management decisions
* Willingness to notify the study staff if they become pregnant during the study
* Willing to sign an informed consent

Exclusion Criteria Summary:

* Currently using a continuous or flash glucose monitoring
* Currently pregnant or planning pregnancy within duration of study or breast feeding; subjects who become pregnant during the study will be withdrawn.
* Conflict of Interest

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
A1c change from baseline after 12 weeks | 12 weeks
  A1c change from baseline after 12 weeks in subjects using new BGMS compared to subjects' pre-study glycemic control

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh, Lothian
  - Highland Diabetes Institute, Inverness

IPD SHARING:
Plan to Share IPD: Yes
Device being used in the study is CE marked and will be used as intended therefore risk is minimal. What? Individual participant data that underlie the results reported in publications, after deidentification (text, tables, figures, and appendices).
  When? Beginning 9 months and ending 36 months following article publication. With whom? Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. For individual participant data meta-analysis. By what mechanism will data be made available? Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available from our archive but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found by reaching out to the study contact listed. What other documents will be available?Abbreviated CSR may be provided upon request and assessment by the company.
Supporting Information: CSR
Time Frame: Up to 12 months post study completion.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.